CLINICAL TRIAL: NCT06044818
Title: Validación Del Sistema de Cribaje y Seguimiento de acceXible Para depresión.
Brief Title: Validation of Accexible as a Tool for Screening and Monitoring Depression.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Accexible (Industry)
Responsible Party: Sponsor
Other Study IDs: PR(AG)86/2023
Record Dates: First submitted 2023-07-13; First posted 2023-09-21 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy
  Interventions: Device: Accexible
- Depression
  Interventions: Device: Accexible

INTERVENTIONS:
Device: Accexible — Speech Analysis

SUMMARY:
Major depressive disorder (MDD) is a chronic disease with a prevalence around 8-12% and is considered one of the most debilitating disease worldwide.

A recent orientation is the analysis of language in relation to the description of images with a high and varied semantic and emotional content. It can be studied that changes in the description of an image check if these changes are associated with the evolution of a person with probable impairment both in memory and cognitive as well as emotional, psychiatric, behavioral and even in their interaction with environmental factors especially those associated with socialization and loneliness.

The present study has the objective of validating Accexible as a tool for Screening and Monitoring Depression.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-65 years of age.
* Participants must have Spanish as their first language (able to speak and understand verbal messages).
* Participants must have mobile phone with internet.
* Participants must have the ability to understand AcceXible's basic instructions.
* Participants must agree to participate in the study and have voluntarily signed the informed consent.

Exclusion Criteria for patients:

* To have received a diagnosis of neurodegeneration.
* To have significant vision problems that would affect the ability to perceive visual stimuli.
* To have significant hearing problems that would affect the ability to understand verbal cues.
* To be unable to give informed consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: adults with suspected depression.
  Controls: healthy controls without depression criteria.
Sampling Method: Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-10-03 (Estimated); Study Completion 2025-01-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Depression | An average of 1 year
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron Institut de Investigación (VHIR), Barcelona, Spain